CLINICAL TRIAL: NCT06692933
Title: Effects of a Hemp Product on the Pharmacokinetics and Pharmacodynamics of Clopidogrel
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Office of Dietary Supplements (ODS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mary Paine, Professor, Washington State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20533; U54AT008909 (NIH)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Interaction
Keywords: CYP2C19; pharmacokinetics; hemp; CBD; natural product; clopidogrel
MeSH Terms: interventions — Cannabidiol; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: clopidogrel alone (Experimental): Participants will be administered a single oral dose (75 mg) of clopidogrel. Blood and urine will be collected for 24 hours.
  Interventions: Drug: Clopidogrel
- Arm 2: chronic hemp (30 mg CBD) + clopidogrel (Experimental): Participants will self-administer a single low dose of hemp (30 mg CBD) as an oral softgel at home daily for 5 consecutive days. On day 6, participants will return to the research setting, where they will be administered a single low dose of hemp (30 mg CBD) and a single oral dose of clopidogrel (75 mg). Blood will be collected for 72 hours and urine will be collected for 24 hours.
  Interventions: Drug: Cannabidiol in the form of hemp; Drug: Clopidogrel
- Arm 3: chronic hemp (240 mg CBD) + clopidogrel (Experimental): Participants will repeat the Arm 2 procedures using a higher dose of hemp (240 mg CBD)
  Interventions: Drug: Cannabidiol in the form of hemp; Drug: Clopidogrel

INTERVENTIONS:
Drug: Cannabidiol in the form of hemp — Cannabidiol (30 mg) in the form of an orally administered hemp oil softgel
  Other Names: CBD
  Arms: Arm 2: chronic hemp (30 mg CBD) + clopidogrel; Arm 3: chronic hemp (240 mg CBD) + clopidogrel
Drug: Clopidogrel — 75 mg oral clopidogrel
  Other Names: Plavix

SUMMARY:
The goal of this clinical trial is to determine how two different doses of cannabidiol (CBD), given as a hemp product, change the blood concentrations of the drug clopidogrel in the body. Results will be used to help design future studies and to assist healthcare providers in informing their patients about the safe use of CBD.

DETAILED DESCRIPTION:
The popularity of cannabis products has grown exponentially over the past decade as several states continue to decriminalize or legalize recreational and/or medicinal use. Cannabis contains >500 phytoconstituents, including >100 cannabinoids. The most well-studied cannabinoids are tetrahydrocannabinol (THC) and cannabidiol (CBD). Although both are psychoactive, THC produces the characteristic "high," while CBD does not. CBD is available as a prescription drug (Epidiolex®) to treat seizure disorders. Hemp, a popular CBD-containing botanical product, is defined as containing <0.3% THC. Hemp was federally legalized in the United States in 2018 following passage of the Farm Bill. Since passage of that bill, hemp and other CBD-containing products have become widely available over the counter. As such, hemp/CBD products have become top-selling botanicals, with sales projected to reach nearly $4.5 billion by 2024. Common uses include self-treatment for pain, anxiety, and sleep disorders.

Despite increasing use of cannabis products, the pharmacokinetic interaction potential with pharmaceutical medications remains understudied. Previous pharmacokinetic studies have yielded convincing evidence that CBD significantly inhibits the activity of the drug metabolizing enzyme cytochrome P450 (CYP) 2C19. Despite the valuable information generated by these and numerous other studies, several unanswered questions about CBD-containing products remain:

1. Do real-world doses and dosing regimens of CBD (< 300 mg) have similar CYP interaction potential as that of higher doses investigated in previous pharmacokinetic studies?
2. What are the effects of CBD on high-impact CYP2C19 substrates, such as the anti-platelet drug clopidogrel (Plavix®)?
3. Does chronic administration of a real-world dose of CBD have similar interaction potential as a very high single dose of CBD?

The primary objective of the proposed study is to evaluate the effects of a well-characterized, widely used hemp product on the pharmacokinetics of the commonly prescribed CYP2C19 substrate clopidogrel (Plavix®) in healthy adult participants who are confirmed to be CYP2C19 normal, rapid, or ultra-rapid metabolizers. Results could be used to inform a future study design involving elderly people, which is a population of interest. Results could also be used to guide healthcare providers in helping their patients make informed decisions about the safe use of hemp

ELIGIBILITY:
Inclusion Criteria:

* 21-64 years old and healthy;
* Confirmed by genetic test to be a CYP2C19 normal, rapid, or ultra-rapid metabolizer;
* Not taking any medications (prescription and non-prescription, including clopidogrel) or dietary supplements/botanical products known to alter the pharmacokinetics of cannabis and/or clopidogrel;
* Have taken hemp or cannabis (in any form) before and tolerated it well;
* Willing to abstain from consuming dietary supplements/botanical products and citrus juices for the duration of the study;
* Willing to abstain from cannabis/marijuana, hemp, THC- and/or CBD-containing products for several weeks;
* Willing to abstain from consuming caffeinated beverages or other caffeine-containing products the evening before and morning of any inpatient day;
* Willing to abstain from consuming alcoholic beverages for one day prior to any inpatient day;
* Willing to use a secondary method of birth control that does not include the introduction or discontinuance of hormonal-based birth control (such as abstinence, copper IUD, or condoms), continuing for 1 week after completing the study;
* Have the ability to and are willing to comply with the requirements of the study;
* Geographically located within a 40-mile radius of Spokane and have the time to participate and;
* Can read and speak English

Exclusion Criteria:

* Under the age of 21 or over the age of 64;
* Any major illness;
* Pregnant or nursing;
* History of allergy or intolerance to cannabis or clopidogrel;
* Taking concomitant medications, both prescription and non-prescription (including clopidogrel) or dietary supplements/botanical products known to alter the pharmacokinetics of cannabis and/or clopidogrel;
* Never taken cannabis (in any form) before;
* Presence of a condition or abnormality that, in the opinion of the Investigator, would compromise participant safety or the quality of the data;
* Currently using or have recently used drugs or other illicit substances for recreational purposes;
* Have used cannabis/marijuana, hemp, THC- and/or CBD-containing products within the last 4 weeks;
* Have an out-of-range clinical laboratory value such that the study physician considers participation in the study a health risk, or;
* Unable to read and speak English

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC ratio of clopidogrel active metabolite | 0-24 hours
  Ratio of the area under the plasma concentration vs. time curve of the active metabolite of clopidogrel in the presence to absence of hemp

SECONDARY OUTCOMES:
Cannabidiol AUC | 0-72 hours
  Area under the plasma concentration vs. time curve of cannabidiol
AUC of cannabidiol metabolites | 0-72 hours
  Area under the plasma concentration vs. time curve of cannabidiol metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University College of Pharmacy and Pharmaceutical Sciences, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication